CLINICAL TRIAL: NCT05667480
Title: Utilization of Immersive Virtual Reality in Computerized Script Training for People with Aphasia: a Feasibility Study
Brief Title: VR and Script Training of PWA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0043271
Record Dates: First submitted 2022-12-11; First posted 2022-12-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-08

CONDITIONS: Aphasia, Acquired; Chronic Stroke
Keywords: functional communication; randomized study; script training; immersive virtual reality; aphasia intervention
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR-based script training (Experimental)
  Interventions: Behavioral: VR-based script training
- Conventional script training (Active Comparator)
  Interventions: Behavioral: Conventional script training

INTERVENTIONS:
Behavioral: VR-based script training — The PWA will wear a head-mounted VR device (e.g., Metaverse Oculus Quest 2 or other commercially available devices) for 30 minutes, which intends to create an immersive environment for training. Scripts trained in the computerized script training program in a particular session will be practiced. Cinematic 360˚ photo-real scenarios of daily contexts such as a restaurant or a grocery store will be displayed in the device while a communication partner, e.g., a waiter in the restaurant or a shopkeeper of a grocery store will initiate the conversation by producing the corresponding part of the script. The PWA will be given time to respond. Upon the completion of PWA's respond, the next conversational turn will be initiated. The clinical assistant, who accompanies the PWA in the entire training session, will control the flow of the 360 ˚ videos.
  Arms: VR-based script training
Behavioral: Conventional script training — The flow of training is identical to the VR condition, except that photos depicting the scenarios and pre-recorded conversational turns will be presented to the PWA on a computer screen with the same procedures mentioned in the VR condition.
  Arms: Conventional script training

SUMMARY:
The goal of this intervention study is to investigate the effects of immersive virtual reality in rehabilitation of language and communication of individuals with post-stroke aphasia. The main research questions are:

1. Is VR-based script training a feasible treatment to Cantonese-speaking PWA?
2. Will VR-based script training, when compared to conventional script training, better enhance treatment outcomes in functional communication of PWA?

Participants will be assessed before, in the middle of, immediately after treatment and 8-week post treatment in terms of their performance on:

1. Accuracy and time for producing trained scripts.
2. Accuracy and time for producing un-trained scripts
3. Standardized aphasia test on severity of language impairment
4. Standardized aphasia test on functional communication

The participants will be randomly allocated to receive one of the treatment:

1. Virtual reality-based computerized script training; or
2. Computerized script training without virtual reality Researchers will compare the treatment outcomes of the two treatment conditions and see if treatment with virtual reality would better promote outcomes when compared to training without virtual reality.

ELIGIBILITY:
Inclusion Criteria:

1. a stroke onset more than six months, with an Aphasia Quotient (AQ) below 96.4, as evaluated by the Cantonese version of Western Aphasia Battery (CAB; Yiu, 1992),
2. premorbid fluent Cantonese speakers,
3. aged between 30 and 80 years,
4. no reported progressive neurogenic disorders such as dementia or Parkinson's disease,
5. no motor speech disorders of moderate to severe level, and
6. normal or corrected-to-normal vision and hearing functions

Exclusion Criteria:

1. concurrent participation in other aphasia treatment trials, and
2. incompatibility with immersive VR exposure such as complains of nausea, headache, or other severe discomforts during trial use of a head-mounted device during screening.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage correct in reading aloud the sentences included in the trained scripts | From baseline up to 1-week post training
  Trained scripts will be shown in written form while the PWA will be asked to read aloud the scripts.
Time required in read aloud of trained scripts | From baseline up to 1-week post training
  Total time to read aloud the trained scripts
Percentage correct in spontaneous production of the sentences included in the trained scripts | From baseline up to 1-week post training
  No written cue will be provided while the PWA will produce the scripts upon questions.
Time required for spantaneous production of trained scripts | From baseline up to 1-week post training
  No written cue will be provided while the PWA will produce the scripts upon questions.

SECONDARY OUTCOMES:
CAB | From baseline up to 1-week post training
  Cantonese version of the Western Aphasia Battery
CANELT | From baseline up to 1-week post training
  Cantonese version of the Amsterdam-Nijmegen Everyday Language Test (ANELT; Blomert et al., 1994)
Percentage correct in producing untrained but related scripts | From baseline up to 1-week post training
  No written cue will be provided while the PWA will produce the untrained scripts that share similar contexts with the trained scripts.

CONTACTS AND LOCATIONS:
Overall Officials: Winsy WS Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, Hong Kong SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The IPD, together with the study protocol, will be shared in an open-access data repository (e.g., Harvard Dataverse).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared starting from three months after manuscript publication.
Access Criteria: The IPD and study protocol will be shared in an open-access data repository without restrictions.